CLINICAL TRIAL: NCT05914389
Title: Induction Chemotherapy Combined With Neoadjuvant Immunotherapy for MSS Colon Cancer: a Prospective Single-center Multi-arm Open-label Randomized Phase II Study
Brief Title: Induction Chemotherapy Combined With Neoadjuvant Immunotherapy for MSS Colon Cancer
Acronym: ICONIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0296
Record Dates: First submitted 2023-05-28; First posted 2023-06-22 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-04

CONDITIONS: Colon Neoplasm
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin; Capecitabine; envafolimab; phosphatidyltransferase, Clostridium butyricum; Colectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard chemotherapy control cohort (Experimental): Patients with locally advanced colon cancer who met the inclusion criteria received two cycles of Capecitabine and Oxaliplatin （Capox） regimen chemotherapy and were evaluated by enhanced CT. Patients with more than 20% regression of maximum diameter of colon tumor in enhanced CT image will be randomly assigned to the Standard chemotherapy control cohort and continued with two more cycles of Capox chemotherapy. Then, these patients will receive curative surgery for colon cancer.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Procedure: Colectomy
- Enhancement regimen of combined Anti-PD-L1 monoclonal antibody (Experimental): Patients with locally advanced colon cancer who met the inclusion criteria received two cycles of Capecitabine and Oxaliplatin （Capox） regimen chemotherapy and were evaluated by enhanced CT. Patients with more than 20% regression of maximum diameter of colon tumor in enhanced CT image will be randomly assigned to the Enhancement regimen of combined Anti-PD-L1 monoclonal antibody and continued with two more cycles of Capox chemotherapy along with the reduced dosage of Anti-PD-L1 monoclonal antibody. Then, these patients will receive curative surgery for colon cancer.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Anti-PD-L1 Monoclonal Antibody; Procedure: Colectomy
- Enhancement regimen of combined lactobacillus and Anti-PD-L1 monoclonal antibody (Experimental): Patients with locally advanced colon cancer who met the inclusion criteria received two cycles of Capecitabine and Oxaliplatin （Capox） regimen chemotherapy and were evaluated by enhanced CT. Patients with more than 20% regression of maximum diameter of colon tumor in enhanced CT image will be randomly assigned to the Enhancement regimen of combined lactobacillus and Anti-PD-L1 monoclonal antibody and continued with two more cycles of Capox chemotherapy along with the reduced dosage of Anti-PD-L1 monoclonal antibody and Clostridium butyricum. Then, these patients will receive curative surgery for colon cancer.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Anti-PD-L1 Monoclonal Antibody; Drug: Clostridium butyricum; Procedure: Colectomy

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 for inducing chemotherapy on Day 1 every 3 weeks and repeat for 4 cycles. The dose reduction protocol for oxaliplatin-induced toxicity was implemented according to the report in BJC (2018) 118:1322-1328.
Drug: Capecitabine — Oral Capecitabine 1000 mg/m2 twice daily combined with oxaliplatin chemotherapy from Day 1 to Day 14 every 3 weeks and repeat for 4 cycles. The dose reduction protocol for capecitabine-induced toxicity was implemented according to the report in BJC (2018) 118:1322-1328.
Drug: Anti-PD-L1 Monoclonal Antibody — The incidence of adverse events with Anti-PD-L1 Monoclonal Antibodies is relatively low. Based on phase I clinical trial data of Envafolimab, a dose reduction design was conducted to minimize the incidence of adverse events while ensuring therapeutic efficacy. In the two cohorts of the efficacy-enhancing design, a reduced dose of 100mg/0.5ml IH QW will be used for 6 weeks. The PD-L1 monoclonal antibody (Envafolimab) dose adjustment was implemented according to the prescribing information.
  Other Names: Envafolimab
  Arms: Enhancement regimen of combined Anti-PD-L1 monoclonal antibody; Enhancement regimen of combined lactobacillus and Anti-PD-L1 monoclonal antibody
Drug: Clostridium butyricum — Clostridium butyricum is treated with Miyarisan 588 powder, 160mg/day (4 packets/day) taken orally for a total of 6 weeks.There have been no reports of adverse reactions for Lactobacillus. There is no predetermined reduction plan.
  Arms: Enhancement regimen of combined lactobacillus and Anti-PD-L1 monoclonal antibody
Procedure: Colectomy — The specific surgical approach, whether it be laparoscopic or open surgery, is determined by the surgeon. The tumor blood supply is ligated and cut at the root of the mesentery, and the margin of resection should be no less than 10cm. Complete resection of the mesocolon (CME) is performed in conjunction.

SUMMARY:
This study aims to elucidate the regression effects of neoadjuvant chemotherapy combined with immunotherapy and adjuvant therapy in locally advanced MSS colon cancer.

DETAILED DESCRIPTION:
The standard treatment for locally advanced colon cancer is surgery followed by adjuvant chemotherapy containing oxaliplatin. The MOSAIC and 16968 studies have shown that approximately 30% of patients experience recurrence and metastasis within 6-7 years after surgery. Neoadjuvant chemotherapy may improve the prognosis of patients with malignant tumors. The significant tumor shrinkage after neoadjuvant therapy indicates a greater likelihood of long-term survival for patients. The OPTICAL and FoxTROT studies have shown that approximately 35% of patients are resistant to oxaliplatin-containing neoadjuvant chemotherapy, with a pCR rate of less than 10% and uncertain survival improvement. In addition, immunotherapy has poor efficacy for microsatellite stable (MSS) patients. Therefore, it is necessary to explore new and effective neoadjuvant treatment modalities for tumor regression.

The study will screen for individuals who are sensitive to oxaliplatin-containing regimens through induction chemotherapy. Immunogenic cell death will be enhanced by oxaliplatin-induced immunogenicity and combined with anti-programmed cell death ligand 1 (PD-L1) monoclonal antibodies for neoadjuvant therapy. In the context of cancer, the role of the intestinal microbiome in mediating immune activation induced by chemotherapy drugs has been demonstrated. Clostridium butyricum will be introduced as an adjuvant to explore the possibility of further increasing the significant response rate of neoadjuvant therapy.

The study will first conduct 2 cycles of Capox induction chemotherapy to screen for patients sensitive to chemotherapy. Patients will be randomized into three cohorts: one chemotherapy standard control cohort (continuing Capox chemotherapy for 2 cycles) and two enhancement design cohorts (Capox chemotherapy + Anti-PD-L1 monoclonal antibody for 2 cycles/Capox chemotherapy + Anti-PD-L1 monoclonal antibody + Clostridium butyricum for 2 cycles), followed by CME surgery. The study's primary endpoint is the proportion of Tumor regression grade(TRG)0/1 in the pathological specimens of surgically resected tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤75 years old.
* Pathologically diagnosed MSS or pMMR-type colon adenocarcinoma.
* The lower edge of the tumor is more than 12cm from the anus as measured by colonoscopy and the lower edge of the tumor cannot be directly palpated during rectal examination.
* Enhanced CT stage T3/4 or T1-4N+ without multiple primary tumors or distant metastasis.
* Life expectancy is expected to be more than 1 year.
* First diagnosis, no previous anti-tumor treatment received, and no chemotherapy contraindications.
* Informed consent, able to understand the study protocol and willing to participate in the study, and will provide written informed consent.

Exclusion Criteria:

* Refused to participate in this study.
* Multifocal colorectal cancer.
* History of malignant tumors, except for basal cell carcinoma, papillary thyroid carcinoma, and various in situ cancers.
* Cannot tolerate chemotherapy, such as but not limited to bone marrow suppression.
* Acute exacerbation of important organ diseases (such as but not limited to COPD, coronary heart disease, and renal insufficiency) and/or severe acute infectious diseases (such as but not limited to hepatitis, pneumonia, and myocarditis), ASA score > 3 points.
* Mental disorders, illiteracy, or language communication barriers that prevent the understanding of the study protocol.
* Tumor obstruction or high risk of obstruction, bleeding, and/or perforation.
* Peripheral sensory neuropathy, unable to receive oxaliplatin-based chemotherapy.
* Pregnancy or lactation.
* Unable to undergo enhanced CT examination or having comorbidities requiring the use of glucocorticoid therapy.
* Continuous use of glucocorticoids for more than 3 days within 1 month prior to signing the informed consent form.
* CT or MRI in the mid-sagittal plane shows that the lower border of the tumor is below the line connecting the sacrococcygeal promontory and the upper border of the pubic symphysis.
* Other situations in which the researcher deems unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
TRG0/1 | 1 day of postoperative pathological examination.
  The sum of tumor regression grades TRG0(disappearance of tumor) and TRG1(scattered residual tumor)(AJCC standard).

SECONDARY OUTCOMES:
AE | Adverse events (NCI CTC AE 5.0) that occurred from the first day of induction chemotherapy to one day before the surgery date(up to half a year).
  the rate of adverse event（AE).
Surgical Complication | From the day of surgery to 30 days after the operation, including intraoperative and postoperative complications.
  the rate of surgical complication during or after operation.
DFS | From date of the patient signs the informed consent form until the date of earliest occurrence of the patient's tumor recurrence or death，whichever came first, assessed up to 36 months.
  3-year Disease-free survival.
OS | From the date of the patient signs the informed consent form until the date of the patient's death, assessed up to 60 months.
  5-year Overall survival.
Concentration of FLT3L | blood tests for FLT3LG at initial diagnosis, after induction chemotherapy, before and 3 months after surgery.
  Fms Related Receptor Tyrosine Kinase 3 Ligand is a marker of immunogenic cell death.
Concentration of cytokines | Blood tests of cytokines such as IFN-γ are conducted using techniques such as immunofluorescence and ELISA at initial diagnosis, after induction chemotherapy, before and 3 months after surgery.
  Blood density measurement of immunoreaction associated cytokines.
T lymphocyte | The types and counts of T cells are analyzed using flow cytometry at initial diagnosis, after induction chemotherapy, before surgery, and 3 months after surgery.
  Cells with cellular immune function.
Molecular pathological analysis of tumor tissue. | Nanostring and Whole exome gene sequencing is performed on tumor specimens to analyze the changes in immune cell types, counts, and other immune status-related factors in the tumor microenvironment before and after treatment (up to half a year).
  Whole exome sequencing and Nanostring to analyze changes in the tumor microenvironment immune status.
Minimal Residual Disease (MRD) | Collect plasma after surgery for MRD detection (up to half a year).
  Minimal Residual Disease which is a potential source of tumor recurrence and distant metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No